CLINICAL TRIAL: NCT02519400
Title: A Single Dose, Double-blind, Genotype-based Stratification Study to Explore the Pharmacokinetics and Pharmacodynamics of Amitriptyline According to CYP2D6 and CYP2C19 Polymorphisms in Healthy Korean Male Adult Subjects
Brief Title: A Genotype Stratification Study for Pharmacokinetics and Pharmacodynamics of Amitriptyline in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyeong-Seok Lim, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PGAM-001
Record Dates: First submitted 2015-08-05; First posted 2015-08-10 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Depression
Keywords: amitriptyline; cyp2d6; cyp2c19
MeSH Terms: conditions — Depression | interventions — Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amitriptyline (Experimental): Single oral dose of amitriptyline, 25 mg
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline — Single oral dosing

SUMMARY:
A total of 24 healthy Korean male subjects will receive a single oral dose of amitriptyline, 25 mg. Subjects will be enrolled in this study based on their cytochrome P450 2D6 and cytochrome P450 2C19 genotypes, and serial blood sampling will be done for plasma concentrations of amitriptyline, nortriptyline, and their metabolites. Various pharmacodynamic markers related to the adverse event of amitriptyline will be measured serially during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age 19~45 years
* The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 28 kg/m2
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial.
* Voluntarily signed the informed consent form

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study
* History of relevant drug allergies or clinically significant hypersensitivity reaction.
* Smoked more than 10 cigarettes a day for past 3 months
* Not eligible due to other reasons including laboratory results

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) of Amitriptyline, 10-Hydroxy-amitriptyline, Nortriptyline, and 10-Hydroxy-nortriptyline | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hour
Maximum concentration (Cmax) of Amitriptyline, 10-Hydroxy-amitriptyline, Nortriptyline, and 10-Hydroxy-nortriptyline | 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hour

CONTACTS AND LOCATIONS:
Overall Officials: Hyeongseok Lim, MD, PhD, Principal Investigator — Asan Medical Center, Ulsan University